CLINICAL TRIAL: NCT04049474
Title: Bronchoscopic Cryo-Immunotherapy of Lung Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00812
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Advanced Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Bronchoscopic Cryo-Immunotherapy (BCI) (Experimental): BCI is performed by advancing a flexible cryoprobe through a bronchoscope to reach a peripheral tumor. The cryoprobe is activated to freeze a portion of the tumor. The cryoprobe is allowed to thaw to prevent removal of lung or airway tissue. The tumor must be located by radial EBUS and a guide sheath placed prior to cryoablation.
  Interventions: Device: ERBOKRYO® CA - Cryosurgical Unit with Flexible ERBECRYO Probe, 1.9 mm outer diameter (ERBE Inc., Tubingen, Germany)

INTERVENTIONS:
Device: ERBOKRYO® CA - Cryosurgical Unit with Flexible ERBECRYO Probe, 1.9 mm outer diameter (ERBE Inc., Tubingen, Germany) — See BCI description.

SUMMARY:
This is a safety and feasibility study of bronchoscopic cryo-immunotherapy (BCI) of peripheral lung tumors in advanced non-small cell lung cancer for the intention of inducing anti-tumor immune responses. The sample size for this study will be 15 patients. Pre- and post- BCI peripheral blood samples will be analyzed to assess for anti-tumor immune responses. Post-BCI peripheral blood will be collected 7 and 14 days after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral lung tumor on pre-procedure chest CT scan, which is known or suspected to be advanced, inoperable non-small cell lung cancer (stages IIIA/B/C and IVA/B) based on the 8th edition TNM staging guidelines
* Pre-procedure chest CT scan with the presence of a bronchus or airway path leading directly to the peripheral lung tumor (also known as a "bronchus sign")
* Undergoing bronchoscopy for diagnostic and/or palliative purpose unrelated to this study.
* Documentation of non-small cell lung cancer either prior to procedure or via on-site pathology review during bronchoscopy (prior to proceeding with planned BCI)
* Ability to provide informed consent
* Concomitant chemotherapy, immunotherapy, and/or radiation therapy are allowed
* ECOG performance status less than or equal to 2

Exclusion Criteria:

* Pregnancy
* Currently on a platelet inhibitor (such as Clopidogrel) other than aspirin or NSAIDS, or on a blood thinner (such as heparin, enoxaparin, or a novel oral anticoagulant), which is unable to be held for planned bronchoscopy
* INR >= 1.5 (post correction)
* Platelets =< 100,000 (post correction)
* Bleeding diathesis
* Contraindication to bronchoscopy
* Absence of tissue diagnosis of non-small cell lung cancer either prior to procedure or during on-site pathology review at time of bronchoscopy.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sterman, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bronchoscopic Cryo-Immunotherapy (BCI)
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bronchoscopic Cryo-Immunotherapy (BCI)
Number analyzed (Participants) | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [61 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Successful Performances Among Patients in Whom BCI is Attempted
Description: Success is defined as identification of the target peripheral lung tumor by radial endobronchial ultrasound within 20 minutes followed by completed cryoablation of target tumor.
Time Frame: Day 0 (Intraoperative)
Measure: Number; unit: Percentage of participants
Arm/Group | Bronchoscopic Cryo-Immunotherapy (BCI)
Number analyzed (Participants) | 21
Percentage of participants | 100

2. Primary Outcome: Percentage of Patients Who Experience Bleeding Complications
Time Frame: Up to Day 7 Post-BCI
Measure: Number; unit: Percentage of participants
Arm/Group | Bronchoscopic Cryo-Immunotherapy (BCI)
Number analyzed (Participants) | 21
Percentage of participants | 0

3. Primary Outcome: Percentage of Participants Who Experience Pneumothorax Requiring Tube Thoracostomy
Time Frame: Up to Day 7 Post-BCI
Measure: Number; unit: Percentage of participants
Arm/Group | Bronchoscopic Cryo-Immunotherapy (BCI)
Number analyzed (Participants) | 21
Percentage of participants | 0

4. Primary Outcome: Length of Time to Perform BCI
Time Frame: Day 0
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Bronchoscopic Cryo-Immunotherapy (BCI)
Number analyzed (Participants) | 21
Seconds | 17 [11.5 to 32.65]

5. Primary Outcome: Length of Fluoroscopy Exposure During BCI
Time Frame: Day 0
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Bronchoscopic Cryo-Immunotherapy (BCI)
Number analyzed (Participants) | 21
Seconds | 201 [135 to 284.5]

6. Primary Outcome: Percentage of Participants Who Experience Grade 4-5 Adverse Events Potentially Related to Procedure
Description: Incidence of National Cancer Institute Common Terminology Criteria for Adverse Events Grade 4 or 5 adverse events that may be possibly, probably, or definitely related to BCI.
Time Frame: Up to Day 7 Post-BCI
Measure: Number; unit: Percentage of participants
Arm/Group | Bronchoscopic Cryo-Immunotherapy (BCI)
Number analyzed (Participants) | 21
Percentage of participants | 0

7. Secondary Outcome: Percentage of Patients With Peripheral Blood CD8+ T Cells Displaying at Least One Combination of Hypothesized Markers
Description: The number of patients whose peripheral blood CD8+ T cells (collected via blood sample) display at least one combination of the following markers after BCI: HLA-DR, CD38, Ki-67, Bcl-2, or PD-1.
Time Frame: Up to Day 14 Post-BCI
Measure: Number; unit: Percentage of participants
Arm/Group | Bronchoscopic Cryo-Immunotherapy (BCI)
Number analyzed (Participants) | 12
Percentage of participants | 50

ADVERSE EVENTS:
Time Frame: 12 months
Description: Systematic - chart review per protocol timelines
Arm/Group | Bronchoscopic Cryo-Immunotherapy (BCI)
All-Cause Mortality (participants affected / at risk) | 3/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT04049474/Prot_SAP_000.pdf